CLINICAL TRIAL: NCT04296487
Title: Introduction of Autologous Chondrocyte Implantation Procedure for the Treatment of Chondral Defect in the Knee
Brief Title: Introduction of ACI for Cartilage Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Dr. Robin Martin, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACI-OTR
Record Dates: First submitted 2019-08-01; First posted 2020-03-05 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Articular Cartilage Defect; Chondral Defect; Osteochondritis
MeSH Terms: conditions — Osteochondritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous Chondrocyte Injection (Experimental): Autologous chondrocytes were isolated and expanded in laboratory, then injected at 2x10^6 of cells per cm^2 of the cartilage defect.
  Interventions: Other: autologous chondrocytes

INTERVENTIONS:
Other: autologous chondrocytes — autologous chondrocytes implantation (ACI)

SUMMARY:
This study was aimed to evaluate effectiveness and safety of autologous chondrocyte suspension for treatment of knee articular cartilage defects.

DETAILED DESCRIPTION:
* Prospective and interventional study
* All procedures are carried out after obtaining informed written consent from patients.
* Study procedures involve a biopsy, cell production, cell implantation and follow-up including a strict post-surgery rehabilitation protocol (12 month timepoint)
* All subjects will be assessed at intervals post-implantation (6 weeks, 3 months, 6 months and 12 months).
* Measures to assess effectiveness and safety will be conducted at follow-ups: Magnetic Resonance Imaging (MOCART score), collection of adverse events, orthopaedic scores (KOOS, IKDC, SF12v2)

ELIGIBILITY:
Inclusion Criteria:

1. Age between 15 and 50.
2. Lesions classified as ICRS Grade III or IV and smaller than 15 cm2
3. Lesions that have failed prior therapy (conservative or surgical treatment ≥ six months)
4. Subjects who understand and sign the consent form for this study

Exclusion Criteria:

1. Body mass index (BMI) of 35 or more
2. Osteoarthritis or rheumatoid arthritis
3. Diffuse lesion
4. Uncorrected mal-alignment, ligamentous instability, or meniscal tear
5. Presence of growth cartilage (15-18 years old)
6. Active smoking or drug consumption
7. Women who are pregnant
8. Positive serology for HIV-1 or HIV-2, Hepatitis B and C and syphilis
9. Proven allergy to porcine collagen, penicillin and gentamicin
10. Poor compliance

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of implantation-associated complications: serious adverse events (SAEs) and serious adverse reactions (SARs) | Up to 12 months.
  Post-implantation data collection: Types, probability and severity of treatment (inflammation, infection,pain, joint effusion, delamination, transplant rejection, fibrocartilage, incomplete cartilage reparation).
Change in tissue integrity into and around the treated aera | 3 months post-implantation
  MRI analysis
Absence of infection after implantation. | 6 weeks post-implantation
  Absence of infection is assessed in blood sample by the quantification of three parameters: C-reactive Protein (CRP), neutrophil and lymphocyte rate. The non-infection is characterised by a CRP rate < 10 mg/L, neutrophil rate ranges from 40-75% and lymphocyte rate ranges from 25-40%.

SECONDARY OUTCOMES:
Self-reported function and knee-related quality of life are assessed by using the Knee injury and Osteoarthritis Outcome Score (KOOS) | Change from baseline to 12 months post-implantation.
  KOOS includes five subscales: symptoms, pain, activities of daily living, function in sport/recreation, and knee-related quality of life. A score in points for each subscale will be calculated, and it ranges from 0 (worst score) to 100 (best score).
Self-reported physical pain and function are assessed by International Knee Documentation Committee score (IKDC) | Change from baseline to 12 months post-implantation
  A score will be calculated, and it ranges from 0 (worst score) to 100 (best score).
Self-reported functional health and weel-being as assessed by SF12 Survey | Change from baseline to 12 months post-implantation
  SF12 survey includes 2 subscales: mental component summary (MCS) and physical component summery (PCS). A score in points for each subscale will be calculated, and it ranges from 0 (worst score) to 100 (best score).
The cartilage repair is assesed by Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) scoring system. | Change from baseline to12 months post-implantation
  MOCART scoring system is based on MRI analysis. A score in points will be calculated, and it ranges from 0 points (no repair) to 100 points (excellent cartilage defect repair)

CONTACTS AND LOCATIONS:
Overall Officials: Robin MARTIN, MD, Principal Investigator — CHUV
Locations (1):
- Centre Hospitalier Universitaire Vaudois - CHUV, Lausanne, Canton of Vaud, Switzerland